CLINICAL TRIAL: NCT05461677
Title: Walking With the SAIRE Smart Walker
Acronym: SAIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Erasmus University Rotterdam (Other); Odisee University College (Unknown)
Responsible Party: Principal Investigator, Ruben Debeuf, Principal investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAIRE Smart Walker
Record Dates: First submitted 2022-07-06; First posted 2022-07-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Gait Disorders in Old Age; Gait Disorders, Neurologic; Walking, Difficulty
MeSH Terms: conditions — Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SAIRE smart walker (Experimental): The investigational device used in this clinical investigation is called the SAIRE smart walker. This first prototype version is equipped with a depth camera and two cheaper cameras. The depth camera is used to acquire high-quality data to train artificial intelligence (AI) models which then can run on the cheaper camera modules. Additionally, two ultrasonic sensors are applied to estimate the distance. A touch monitor is used to provide audiovisual feedback and display the user interface. Two LED strips are also attached to the walker to provide additional visual feedback to the patient.
  The SAIRE smart walker gives feedback to the patient in terms of cadence using a metronome, and foot placement using the LED strips and the video stream presented on the monitor. Additionally, the walker will give information about step length and step width through AI-models.
  Interventions: Device: SAIRE smart walker
- Standard walker (Active Comparator): The comparator device consist of a standard 4-wheeled walker
  Interventions: Device: Standard 4-wheeled walker
- No walking aid (Active Comparator)
  Interventions: Other: No walking aid

INTERVENTIONS:
Device: SAIRE smart walker — Participants will walk along the 10-meter walkway 5 times using the SAIRE smart walker
  Arms: SAIRE smart walker
Device: Standard 4-wheeled walker — Participants will walk along the 10-meter walkway 5 times using a standard 4-wheeled walker
  Arms: Standard walker
Other: No walking aid — Participants will walk along the 10-meter walkway 5 times without using a walking aid
  Arms: No walking aid

SUMMARY:
The current study aims to investigate the effect of walking with the SAIRE smart walker on spatiotemporal parameters and gait kinematics in a population who suffer from difficulties during gait, and compare this to walking with a standard walker or no walking aid.

DETAILED DESCRIPTION:
This study is an experimental single group study investigating the effect of walking with a smart walker compared to walking with a standard walker or no walking aid in persons who suffer from gait difficulties. Participants will perform one session of walking in three different conditions, (1) walking with the SAIRE smart walker, (2) walking with a standard walker and (3) if the participants are able to walk without the use of an assistive device, walking without a walker. During this session, gait parameters will be compared between the three conditions.

Experimental session: During the experimental session, participants will walk along the 10-meter walkway (5 times for every condition) After every 5 trials, a rest period of minimum 5 minutes will be held to avoid fatigue. Three different walking conditions will be measured: (1) walking with the SAIRE smart walker, (2) walking with a standard walker and if possible (3) walking with no walking aid. Each walking condition will be measured five consecutive times in a randomized order. The order of the conditions will be randomized using closed envelopes containing notes that say what order of conditions will be used. This randomization is done to avoid fatigue effects that might occur when a strict order is used.

Before the start of the experimental session, participants will practice using the SAIRE smart walker for maximum 10 minutes to familiarize with the feedback given by the walker. After this familiarization session, the surface electrodes and reflective markers will be placed on the participants and the experimental session will start.

Analysis: This study will investigate the difference in gait biomechanics of adults with gait difficulties while using different walking aids.

Descriptive statistics of the baseline characteristics of all participants will be performed. The effect of gait with a smart walker on spatiotemporal gait parameters, kinematics and muscle activity will be compared to gait with a standard 2-wheeled walker and gait without a walking aid. Data will be visualized using LO(W)ESS smoothing (locally weighted scatterplot smoothing) to explore the effect (per condition and outcome). Values will be compared between conditions in a one-way repeated measures analysis of variance. For the analysis of the USE questionnaire, percentage distribution of every item and mean scores for every subscale will be calculated using Microsoft Excel (Microsoft, Washington, DC).

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk along a 10-meter walkway multiple times over a period of 120 minutes
* Ambulation with any sort of assistive device (e.g. cane, crutches, walker, etc.)
* Sufficient arm/hand function to walk with a walker
* Capable of understanding and carrying out instructions
* Capable of giving informed consent

Exclusion Criteria:

* Presence of cognitive impairement (MoCA score <23)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
3D kinematic measurements of the lower limb | At the end of the experimental session, Day 1
  Kinematic data (i.e., movement amplitudes of the bilateral hip, knee and ankle joint) of the lower limbs during walking will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Walking speed | At the end of the experimental session, Day 1
  Walking speed will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Cadence | At the end of the experimental session, Day 1
  Cadence will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Step length | At the end of the experimental session, Day 1
  Step length will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Step time | At the end of the experimental session, Day 1
  Step time will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Swing time of the lower limbs | At the end of the experimental session, Day 1
  Swing time of the lower limbs during walking will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Stance time | At the end of the experimental session, Day 1
  Stance time of the lower limbs during walking will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Single limb support period | At the end of the experimental session, Day 1
  Single limb support period will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Double limb support period | At the end of the experimental session, Day 1
  Double limb support period will be recorded continuously with the use of a 14-camera Vicon Vero 1.3 system at 100 Hz.
Electromyography | At the end of the experimental session, Day 1
  Muscle activity of the lower limb muscles (bilateral: M. rectus femoris, M. vastus lateralis, M. biceps femoris, M. tibialis anterior, M. gastrocnemius medialis) will be recorded continuously during treadmill walking with the use of surface electrodes. Signals will be recorded with the wireless Cometa Wave Plus EMG system (16 channels).

SECONDARY OUTCOMES:
User experience with a modified version of the USE questionnaire | At the end of the experimental session, Day 1
  User experience will be assessed using a translated version of the self-administered Usefulness, Satisfaction and Ease of use (USE) questionnaire. This scale ranges from 30 to 210, with a higher score translating to higher satisfaction. Additionally, open questions were added to the questionnaire to uncover possible barriers and facilitators in the use of the smart walker.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Swinnen, Prof. Ph.D, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Brubotics Rehabilitation Research center, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No